CLINICAL TRIAL: NCT07400458
Title: Long-term Follow-up Study Following the Approval of Hearticellgram-AMI Administration to Evaluate Its Safety in Patients With Acute Myocardial Infarction
Brief Title: Long-term Follow-up Study Following the Approval of Hearticellgram-AMI Administration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PMC-P-13
Record Dates: First submitted 2024-05-09; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hearticellgram-AMI (Experimental): Patients with Acute Myocardial Infarction who had administered Hearticellgram-AMI.
  Interventions: Biological: Hearticellgram-AMI

INTERVENTIONS:
Biological: Hearticellgram-AMI — Patients who had administered Hearticellgram-AMI.

SUMMARY:
This Long-term follow-up is designed to evaluate the safety of patient with Acute Myocardial Infarction who had administered Hearticellgram-AMI.

DETAILED DESCRIPTION:
To evaluate the safety for 60 months after a single dose of Hearticellgram-AMI in patients with Acute Myocardial Infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Those who had administered Hearticellgram-AMI
2. Those who voluntarily agreed in writing to participate in this investigation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2028-10-12 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of AESI | For 5 years
  death, neoplasms or malignancies in tissues or organs, Immune response

CONTACTS AND LOCATIONS:
Locations (1):
- KIMHYUNSOO Clinic, Seoul, Gangnam, South Korea